CLINICAL TRIAL: NCT01939886
Title: Treatment Efficacy and Malaria TRANSmission After Artemisinin Combination Therapy 2 (TRANSACT2)
Acronym: TRANSACT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Radboud University Medical Center (Other); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRANSACT 2
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Malaria
Keywords: Malaria treatment efficacy; Malaria transmission
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemether- Lumefantrine (Experimental): Treatment with artemether-lumefantrine (AL; Coartem; Novartis Pharma), administered as half a tablet (20 mg of artemether and 120 mg of lumefantrine) per 5 kg of body weight in a 6-dose regimen (at enrolment and 8, 20, 32, 44, and 56 h [+/-90 min] after the initiation of treatment). AL is currently the first line treatment in Tanzania Other Name: Coartem;
  Interventions: Drug: Artemether-lumefantrine combination
- Drug: Mefloquine-Artesunate, an alternative ACT (Active Comparator): Treatment with the paediatric fixed dose combination Mefloquine-Artesunate (MQ-AS; Artequin; Mepha, Aesch, Basel, Switzerland, artesunate (50 mg/day) and mefloquine (125 mg/day) fixed dose formulation (stick pack) once daily for 3 consecutive days, given in three daily doses. The weight range of enrolled children is chosen to be recommended for this fixed dose combination. MQ-AS is available in Kenya as Artequin and has been extensively tested in uncomplicated malaria in children.
  Interventions: Drug: Mefloquine - Artesunate

INTERVENTIONS:
Drug: Mefloquine - Artesunate
  Other Names: Artequin
  Arms: Drug: Mefloquine-Artesunate, an alternative ACT
Drug: Artemether-lumefantrine combination
  Other Names: Coartem
  Arms: Artemether- Lumefantrine

SUMMARY:
Artemisinin combination therapy (ACT) with artemether lumefantrine (AL) is currently the first line treatment policy in Kenya. AL is an efficacious drug that also has the capacity to reduce malaria transmission to mosquitoes. Nevertheless, there is concern about the development of parasite resistance against AL. Clinical trials in Asia showed that mefloquine-artesunate (MQ-AS) may be more efficacious than AL and may have a more pronounced beneficial effect on post-treatment malaria transmission. MQ-AS is registered and used in Kenya but there have been no reported direct comparisons of AL and MQ-AS with clinical and transmission endpoints (i.e. adequately clearing parasites and preventing transmission to mosquitoes).

Screening for molecular markers that are related to parasite susceptibility to ACT drugs and to post-ACT treatment malaria transmission can assist strategies to prevent the development and spread of ACT resistance.

In the current study, we compare AL and MQ-AS for the treatment of uncomplicated malaria. Our endpoints are i) clinical efficacy, ii) post-treatment gametocytaemia by molecular techniques.

In the current study, the investigators compare AL and MQ-AS for the treatment of uncomplicated malaria. The investigators endpoints are

clinical efficacy post-treatment gametocytaemia by molecular techniques

DETAILED DESCRIPTION:
Accurate diagnosis followed by prompt and efficacious treatment is the backbone of any malaria control programme. However, malaria treatment has been facing huge challenges in recent years. A number of affordable antimalarial drugs have been used to cure malaria since the 1940s: these include chloroquine (CQ), sulphadoxine-pyrimethamine (SP; Fansidar®), mefloquine (MQ), amodiaquine (AQ) and quinine. The emergence and spread of resistance to these commonly-used drugs has been largely responsible for the worsening of the malaria situation observed in the past decades.

Across the African continent, guidelines have recently been changed. The World Health Organization (WHO) recommends for falciparum malaria the use of combination therapies, preferably those containing artemisinin derivatives (ACT, artemisinin-based combination therapy). Artemisinin derivatives, e.g. artesunate, artemether and dihydroartemisinin, being extremely potent antimalarial agents are the ideal partners in combinations with other antimalarials. ACTs have three demonstrable advantages over conventional therapy, they i) are efficacious in clearing asexual parasites, ii) substantially reduce post-treatment gametocyte carriage and iii) "protect" the partner drug from selecting resistant parasites.

In Kenya, both CQ and SP have lost clinical efficacy. CQ was replaced by SP in 1998 and in the year 2006, SP was effectively replaced by Artemether-Lumefantrine (AL: Coartem®). The policy change to the artemisinin-based drug AL is in line with the WHO recommendations to shift to ACT as first line antimalarial treatment.The most efficacious ACT, however, needs local comparisons in terms of treatment efficacy and transmission-reducing activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 10 years
* Residents of research area (5 km around the clinic)
* Willingness to come for complete scheduled follow-up.
* Uncomplicated malaria with P. falciparum mono-infection
* Parasitaemia of 1000-200,000 parasites/ul
* Temperature > 37.5°C and < 39.5°C, or history of fever in previous 24 hours.
* No history of adverse reactions to AL
* Understanding of the procedures of the study by parent or guardian and willing to participate by signing informed consent forms.

Exclusion Criteria:

* General signs of severe malaria
* Haemoglobin concentration < 5g/dl
* Presence of disease other than malaria causing febrile conditions
* Mixed infection with P. malariae or other non-falciparum malaria species
* Unwilling to participate and sign informed consent forms.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the number of participants with clinical and parasitological treatment failure after treatment artemether-lumefantrine (AL) and mefloquine-artesunate MQ-AS | 42 day follow-up
  Parasite prevalence will be determined by microscopy and molecular methods on days 3-42 after intitiation of treatment. Clinical (fever+parasitological failure) and parasitological efficacy will be determined in relation to treatment arm and parasite clearance dynamics

SECONDARY OUTCOMES:
the number of individuals with gametocytes after treatment with AL or MQ-AS | 42 days follow-up
  gametocyte carriage will be determined by microscopy and molecular QT-NASBA to generate gametocyte prevalence estimates on follow-up days and the mean duration of gametocyte carriage in days.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sawa, MB.Ch.B, MSc., Principal Investigator — KCMC/ICIPE; Jaffu Chilongola, PhD, Principal Investigator — KCMC; Colin Sutherland, PhD, Study Director — London School of Hygiene and Tropical Medicine; Henk Schallig, PhD, Study Chair — KIT, Amsterdam
Locations (1):
- St. Jude's Clinic, ICIPE Thomas Odhiambo Campus, Mbita, Nyanza, Kenya

REFERENCES:
- [Background] Beshir KB, Sutherland CJ, Sawa P, Drakeley CJ, Okell L, Mweresa CK, Omar SA, Shekalaghe SA, Kaur H, Ndaro A, Chilongola J, Schallig HD, Sauerwein RW, Hallett RL, Bousema T. Residual Plasmodium falciparum parasitemia in Kenyan children after artemisinin-combination therapy is associated with increased transmission to mosquitoes and parasite recurrence. J Infect Dis. 2013 Dec 15;208(12):2017-24. doi: 10.1093/infdis/jit431. Epub 2013 Aug 14. PMID 23945376
- [Background] Sawa P, Shekalaghe SA, Drakeley CJ, Sutherland CJ, Mweresa CK, Baidjoe AY, Manjurano A, Kavishe RA, Beshir KB, Yussuf RU, Omar SA, Hermsen CC, Okell L, Schallig HD, Sauerwein RW, Hallett RL, Bousema T. Malaria transmission after artemether-lumefantrine and dihydroartemisinin-piperaquine: a randomized trial. J Infect Dis. 2013 Jun 1;207(11):1637-45. doi: 10.1093/infdis/jit077. Epub 2013 Mar 6. PMID 23468056